CLINICAL TRIAL: NCT06619379
Title: The Effect of Vaginal Speculum Type and Retention Time on Pregnancy Outcomes During The Embryo Transfer Process
Acronym: Speculum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofertil IVF Health Center (Other)
Responsible Party: Principal Investigator, Elif Güler Ergin, MD, Embryologist, Eurofertil IVF Health Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Eurofertil
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Rates
Keywords: IVF embryo transfer speculum retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plastic speculum (Other): Metal speculum
  Interventions: Other: Retention time of speculum
- Metal speculum (Other): Metal speculum will be used in this group
  Interventions: Other: Retention time of speculum

INTERVENTIONS:
Other: Retention time of speculum — According to the randomization, the speculum can be extracted :
  1. just after the transfer catheter is withdrawn
  2. 60 seconds after the transfer catheter is withdrawn
  3. 420 second (7 minutes) after the catheter is withdrawn

SUMMARY:
Investigators aim to investigate possible affects of a speculum material and retention strategy on IVF pregnancy results. The study is planned as a prospective, randomized control trial. All of the clinical managements, including the embryo transfers, will be performed by the same gynecologist for homogeneity of the study. Only the cases with good implantation potentials are going to be included. Therefore, transfers with cleavage embryos and blastocysts rather than good and top quality will be excluded. All patients included to final statistical analysis will receive the same luteal support.

DETAILED DESCRIPTION:
Participants will be included among the 20 - 40 years old women applying to for IVF. Women with mullerian anomalies and couples with chromosomal abnormalities will be excluded. Histrory of recurrent implantation failure, thin endometrium will also be considered as exclusion criterias. Participants who are initially included in the study will be excluded either the demanded preimplantation genetik testing for aneuploidy optionally, or if the embryo transfer is performed under general anesthesia or the embryo transfer is recorded as difficult transfer.

The participants included in the study will be randomised for the speculum material ( metal or plastic) and also for the retention time of the speculum out of the vagina. Just immediately before applying the speculum to the patient, the material temperature will be measured and recorded with a thermometer capable of digital and object measurement.

All of the transfers will be performed with the same technique. After the embryo transfer is made and the transfer catheter is withdrawn, the speculum will be extracted according to the randomization. If the speculum is not extracted immediately, the chronometer will be started and the extraction will be done either in the 60. second or 420. second ( 7 minutes) according to the randomization . As there are two speculum materials and three retention time arms in the design, a total of 6 groups will be formed after crossover. Data gained in this way will be analyzed and their demographic data and embryological parameters will be evaluated and the implantation rates, pregnancy rates and clinical pregnancy rates of the patients will be determined.

ELIGIBILITY:
Inclusion Criteria:

* women aged 20-40
* cases that good and top quality embryos are achieved for embryo trasnfer

Exclusion Criteria:

* recurrent implantation failure
* any known genetic problems of couple
* any known mullein anomalies
* PGT-A cases
* thin endometrium

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — the participants are women whom embryo transfer will be performed
Enrollment: 200 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pregnacy rates | Beta-HCG test will be taken on the 12th day of the embryo transfer
  Pregnancy rates is the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofertil, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Without sharing the names of the participants, additional data can be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available after the study is submitted to a journal. There is not a limitation for the duration of availability
Access Criteria: The reviewers can be able access the IPD and supporting information. Requests by email will be acceptable for data rather than names of participants